CLINICAL TRIAL: NCT04815057
Title: The Effects of Wellness Education Given to 5th Grade Students During the Covid-19 Pandemic Process on Their Quality of Life and Physical Activity
Brief Title: The Effects of Wellness Training Given to Fifth Grade Students During the Covid-19 Epidemic Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sumeyra Yılmaz (Other)
Responsible Party: Sponsor-Investigator, Sumeyra Yılmaz, Responsible investigator, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Sağlık Bilimleri Univesity
Record Dates: First submitted 2021-03-11; First posted 2021-03-24 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Health Behavior
Keywords: wellness; adolescent; quality of life; physical activity
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Masking Description: the researchers evaluating the outcomes were blinded in determining the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Experimental): wellness education
  Interventions: Behavioral: Wellness Education

INTERVENTIONS:
Behavioral: Wellness Education — The wellness education given to fifth grade students and the quality of life, its effect on physical activity status

SUMMARY:
This study conducted an experimental study with a randomized control group to decide on the quality of life and physical activity of the Wellness education for fifth grade students during the Covid-19 pandemic process.

DETAILED DESCRIPTION:
After the population and sample calculations were made, the students who had their pre-tests were randomized to the Wellness Education Group and the Control Group. In this study conducted in two state secondary schools affiliated to Kırşehir Provincial Directorate of National Education, the experimental group was given Wellness training. No intervention was made to the control group. Four weeks after the training, the students were post-tested and the data were analyzed.

In order not to affect the groups from the practices to be made, first of all, schools were randomized and the schools were divided into Wellness Education Group and Control Group with a closed envelope lot method. Prof. Dr. Erol Güngör Secondary School (Group I) Wellness Education Group has been assigned to Kırşehir Merkez Yunus Emre Secondary School (Group II) Control Group. Experimental and control groups in order to reduce selection bias and control variables that may have an effect on outcome variables; A randomized assignment was made by a statistician who did not know the names and characteristics of the students. In determining the students to be included in the study; Student lists and the Excel 2016 program were used, and Simple Random Sampling was performed. The student lists assigned to the groups by the expert were submitted to the researcher before the initiatives started.

ELIGIBILITY:
Inclusion Criteria:

* Being a fifth grade student,
* Not having any physical or mental disability,
* Agree to participate in research,
* Not allowed to participate in research by their parents.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Turkish child physical activity questionnaire | 3month
  The predictive self-report gazelle is a seven-day recall scale to assess mid-to-high physical activity in children aged -14 years. Calculation of the total score of the questionnaire; The score obtained after adding the scores of the answers to the questions 1, 2, 3, 4, 5, 6, 7, 8, and 9 and dividing by the number of questions is the total physical activity score of the child from the questionnaire.
  It is conducted on a 5-point scale for each item of the questionnaire and has a score between 1-5. "1" indicates low physical activity, "5" indicates high physical activity. A high score means good physical activity.

SECONDARY OUTCOMES:
quality of life scale for children | 3 month
  quality of life score of students will increase after education, Items score between 0 and 100. Never 100 points, rarely He gets 75 points, sometimes 50 points, often 25 points and almost always 0 points. 5-7 years old child In his form he never gets 100 points, sometimes 50 points and often 0 points. Taken from substances The total score of the scale is obtained by dividing the scores by the number of filled items., high score means good quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Second School, Kırşehir, Turkey (Türkiye)